CLINICAL TRIAL: NCT06002867
Title: Investigation of the Effect of Serratus Anterior Plan Block on Postoperative Pain in Patients Who Underwent Minimally Invasive Cardiac Surgery.
Brief Title: Serratus Anterior Plan Block and Postoperative Pain in Patients Who Underwent Minimally Invasive Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Yavuz Orak, Associate professor, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2022/16-03
Record Dates: First submitted 2023-05-31; First posted 2023-08-21 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Morphine Consumption; Pain
Keywords: Serratus anterior plan block; Postoperative Pain; Minimally Invasive Cardiac Surgery
MeSH Terms: conditions — Pain; Pain, Postoperative | interventions — Saposins; Dental Occlusion

STUDY DESIGN:
Intervention Model Description: Grup SAPB
  Grup Control
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group SAPB (Serratus anterior plane block) (Active Comparator): Active Comparator: Group SAPB (Serratus anterior plane block) After the operation is completed, the block operation will be performed while intubated. The patient will be in the supine position.
  The area where the procedure will be performed will be cleaned with povidone iodine.
  The latissimus dorsi muscle and the serratus muscle will be visualized at the level of the 4th and 5th ribs using a 22-gauge, 80 mm insulated Quincke type needle with the 'in plane' technique, accompanied by a high frequency (10-18 MHz) ultrasound linear probe covered with a sterile sheath. .
  After the fascia between the two muscles is fixed, the block needle will be advanced from caudal to cranial and 40 ml (20 ml local anesthetic + 20 ml saline) 0.25% local anesthetic will be injected on the serratus muscle between the two muscles.
  Interventions: Procedure: SAPB (Serratus Anterior Plan) Block
- Group Control (No Intervention): The action will not be applied

INTERVENTIONS:
Procedure: SAPB (Serratus Anterior Plan) Block — The patient will be in the supine position. The area where the procedure will be performed will be cleaned with povidone iodine. Using a 22-gauge, 80 mm insulated Quincke needle with a high frequency (10-18 MHz) ultrasound linear probe covered with a sterile sheath, the latissimus dorsi muscle and the serratus muscle will be visualized at the level of the 4th and 5th ribs. After determining the fascia between the two muscles, the block needle will be advanced from caudal to cranial and 40 ml of 0.25% bupivacaine (local anesthetic) will be injected on the serratus muscle between the two muscles.
  Arms: Group SAPB (Serratus anterior plane block)

SUMMARY:
Acute postoperative pain is defined as sudden onset pain that develops after stimulation due to surgical intervention. It is most severe in the first 24 hours after surgery and gradually decreases in severity and creates dissatisfaction in the patient. Postoperative pain that cannot be treated properly can cause various systemic effects, prolongation of hospital stay, decrease in patients' quality of life, and development of chronic pain. An increase in blood pressure, heart rate, cardiac irritability and systemic vascular resistance is observed with the sympathetic response due to pain. Increased myocardial workload and oxygen consumption may increase or trigger myocardial ischemia. Pulmonary dysfunction has an important place in the determination of mortality and morbidity after surgery and anesthesia.Especially in patients who have undergone thoracic surgery, pain limits the movements of the thoracic muscles, reducing functional residual capacity and vital capacity.This causes the development of atelectasis in the patient and the development of hypoxia and pneumonia due to the deterioration of the ventilation/perfusion ratio. Effective analgesia can be achieved in the postoperative period by administering a certain volume of local anesthetic between any two muscle planes using USG. In SAPB, a local anesthetic is injected between the serratus anterior muscle and the latissimus dorsi muscle to create sensory paresthesia in the thoracic wall. It is known to reduce pain scores in the postoperative period.

Serratus anterior plane block is a safe facial plane block performed under USG guidance.Depending on the application site of the block and the amount of local anesthetic administered, different numbers of intercostal nerves, long thoracic nerves and thoracodorsal nerves may be affected. The fact that Serratus anterior plane block (SAPB) is effective between T2-T9 dermatomes enables it to be used effectively in lateral thoracic wall surgeries.

DETAILED DESCRIPTION:
Patients between the ages of 18-65 who will undergo minimally invasive cardiac surgery under elective conditions will be included in the study.

Patients will be randomized. The patients will be included in the study after they are informed about the study and their consent is obtained with the patient consent form. Patient groups will be divided into two groups as SAPB Group (n=20) and Control Group (n=20). All patients will be intubated with a double lumen endotracheal intubation tube in accordance with general anesthesia rules. Patients' age, weight, height, body mass index (BMI), additional disease, surgery, medications used, Ejection/Fraction, platelet count (x10/L), cardiopulmonary bypass time (min), aortic cross clamp time (min) , intraoperative remifentanil amount (mcq), intraoperative morphine dose (0.1 mg/kg), postoperative extubation time (min), post extubation, 1. hour, 2nd hour, 4th hour, 8th hour, 12th hour, 24th hour NRS (Numerical Rating Scale) pain score (between 0 and 10, no pain at 0, maximum pain at 10), extubation after, 1st hour, 2nd hour, 4th hour, 8th hour, 12th hour, 24th hour morphine consumption (Patient Controlled Analgesia), how many additional doses paracetamol was administered, how many additional doses were administered, additional analgesic need time (minutes), postoperative hemodynamic monitoring, 1st hour, 2nd hour, 4th hour, 8th hour, 12th hour, 24th hour PH, PO2 (oxygen pressure) ), MAP (mean arterial pressure), will be recorded. In addition, nausea, vomiting, itching, constipation, and the duration of intensive care hospitalization will also be recorded in the postoperative period. The patient will be told to express the degree of postoperative pain using the numerical scoring scale (NRS) before the operation. The patient will be informed about the PCA to be inserted in the postoperative period. After the surgical procedure is completed, serratus anterior plane block will be applied to the patients under the guidance of postoperative USG. After the surgery, the patients will be transferred to the cardiovascular surgery intensive care unit.

Serratus Anterior Plan (SAP) Block:

After the operation is completed, the block operation will be performed while intubated. The patient will be in the supine position.

The area where the procedure will be performed will be cleaned with povidone iodine. With a high frequency (10-18 MHz) ultrasound linear probe covered with a sterile sheath, using the 'in plane' technique using a 22-gauge, 80 mm insulated Quincke type needle, midaxillary line with the latissimus dorsi muscle and serratus at the level of the 4th and 5th ribs. After determining the fascia between the two muscles by imaging the muscle, the block needle will be advanced from caudal to cranial and 40 ml of 0.25% bupivacaine will be injected on the serratus muscle between the two muscles. No block will be applied to the control group. Only the PCA (Patient Control Analgesia) drug with Morphine will be used.

In the intensive care unit, the patients will be extubated after respiratory effort appears, when the patient is awake, blood gas values are within the normal range, body temperature is normal, and hemodynamically stable. When NRS is >3-4, patients will be instructed to press the PCA device. If the patient's consciousness and hemodynamic status do not allow for pain assessment, the patient will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-65,
* Coronary artery patients with normal left ventricular function and scheduled for elective coronary artery bypass surgery,
* Valve diseases for which elective valve replacement is planned with normal left ventricular function,
* Cases of ASD (Atrial Septal Defect) for atrial septal defect closure
* Patients who will have elective valve + coronary artery bypass without left ventricular dysfunction and patients who volunteer to participate in the study,
* No coagulation disorder
* Patients with a platelet count of more than 100,000,
* Patients with good mental status,
* Patients with an ejection difference value (E/F) above 50% will be included in the study.

Exclusion Criteria:

* Cases that will require emergency and repeat heart surgery,
* With advanced left coronary artery disease and left ventricular dysfunction,
* Receiving preoperative inotropic support therapy for any reason,
* Mitral stenosis with atrial thrombus,
* Patients with low cardiac out put syndrome and E/F below 50%,
* Patients who need intra-aortic balloon pump during surgery,
* Patients with bleeding and coagulation disorders,
* Patients with hepatic and renal dysfunction,
* Patients with Uncontrolled Diabetes Mellitus and Chronic Obstructive Pulmonary Disease,
* Patients allergic to opioids, analgesics and bupivacaine,
* Patients with atrial fibrillation using anticoagulants,
* Patients with cognitive dysfunction
* Patients who do not want to participate in the study will be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-04-10 (Actual)

PRIMARY OUTCOMES:
Morphine consumption by PCA (Patient Control Analgesia) | The change from baseline in the postoperative period at the 1, 2, 4, 8, 12 and 24th hour after extubation
  Morphine consumption used in case of pain

SECONDARY OUTCOMES:
pain (NRS)score | Change from baseline of NRS Score at 1,2, 4,,8, 12 and 24 hours after being extubated will be recorded.
  Change from baseline NRS Score. from 1 to 10 , 0: No pain, 10: 10 pain that can not be
PH | Change from baseline of PH at the 1, 2, 4, 8, 12 and 24th hour after extubation
  PH change after extubation
PO2 | Change from baseline of PO2 at the 1, 2,4 , 8, 12 and 24th hour after extubation
  PO2 change after extubation
Mean Arterial Pressure (MAP) | Change from baseline of MAP at the 1, 2, 4, 8, 12 and 24th hour after extubation
  MAP change after extubation
PCO2 | Change from baseline of PCO2 change at the 1, 2, 4, 8, 12 and 24th hour after extubation
  PCO2 change after extubation

CONTACTS AND LOCATIONS:
Overall Officials: Yavuz Orak, Principal Investigator — Kahramanmaraş Sütçü İmam Üniversitesi Tıp Fakültesi, Anesteziyoloji ve Reanimasyon Bölümü
Locations (1):
- Kahramanmaras Sutcu Imam University Faculty of Medicine, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No